CLINICAL TRIAL: NCT01688388
Title: Single Fraction Intraoperative Radiotherapy With Electrons: An Option in Breast-Conserving Operable Breast Cancer Stages 0, I and II - Prospective, Single-arm Trial
Brief Title: Single Fraction Intraoperative Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph Hospital of Orange (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-001 Single Fraction IORT
Record Dates: First submitted 2012-09-12; First posted 2012-09-19 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Invasive Ductal and Invasive Lobular Breast Carcinoma; Stage 0 Breast Carcinoma; Stage I Breast Carcinoma; Stage II Breast Carcinoma
Keywords: Breast Cancer; Carcinoma; Radiotherapy; Intraoperative Radiotherapy; IORT
MeSH Terms: conditions — Carcinoma, Lobular; Breast Carcinoma In Situ; Breast Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IORT Arm (Experimental): Intraoperative radiotherapy (IORT) is delivered after completion of the lumpectomy and sentinel node procedure.
  Interventions: Procedure: Intraoperative Radiotherapy

INTERVENTIONS:
Procedure: Intraoperative Radiotherapy — Intraoperative radiotherapy (IORT) is delivered after completion of the lumpectomy and sentinel node procedure. IORT is performed on mobile or fixed linacs with variable electron energies in the range of 6-12 MeV prescribed to a dose of 21 Gy, with the prescription dose covering at least 90% of the Planning Target Volume (PTV). PTV is defined as a 3D volume of 1-2 cm beyond the former macroscopic tumor edge (excluding skin, limit to anterior rib surface: 5 Gy). The choice of electron energy as well as the cone applicator size has to account for minimum PTV requirements. Tissue depth measurement will be documented by intraoperative sonography.
  Other Names: IORT

SUMMARY:
This clinical trial is being conducted to find out the effects (good and bad) of giving the full radiation treatment for breast cancer as a single dose of radiation during surgery for breast cancer. This single fraction intraoperative radiotherapy with electrons will study the toxicity, local control and cosmetic outcome.

DETAILED DESCRIPTION:
For patients with certain types of breast cancer, one standard treatment is breast conserving surgery or lumpectomy (surgery to remove abnormal tissue or cancer from the breast and a small amount of normal tissue around it) followed by breast radiation. The radiation treatment in this situation usually lasts 3 to 5 1/2 weeks followed by 5-8 daily localized irradiation (or boost) treatments at the site where the lump was removed. During this study, the single dose of electron irradiation given at the surgical site during the operation will replace the radiation given after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven invasive breast carcinoma ductal, lobular and/or Ductal Carcinoma in situ
* Age > 40 years
* Karnofsky performance status > 70%
* Tumor. Single discrete tumor or focal microcalcifications that can be imaged on a specimen radiograph or multifocal disease within the same quadrant with a maximum dimension of equal to or less than 2.5 cm
* Nodal Status: preoperatively N0
* Clear surgical margins: R0
* All grades G1 - G3
* Any hormonal receptor and HER-2 status
* Informed consent

Exclusion Criteria:

* Gender: male
* Tumor size: more than 2.5 cm
* Nodal status greater than or equal to N1 pathologically
* Multicentricity
* Previous radiotherapy to the involved breast
* Karnofsky Index < 70%
* Mixed connective tissue diseases e.g. rheumatoid poly arthritis, thromboangitis obliterans, systemic lupus
* Distant metastases
* Pregnancy in woman of child bearing age
* Unable to provide written consent

Ages: 41 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-02; Primary Completion 2016-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Toxicity Assessment | 5 years
  Assessment of acute toxicity of breast irradiation according to CTC-toxicity Scoring - system:
  * End of initial surgical phase: Week 1, 4
  * First Follow-up investigation: Month 2 Assessment of late toxicity according to NSABP scoring-systems at 6, 12, 24, 36, 48, and 60 months

SECONDARY OUTCOMES:
Cosmetic Evaluation | 5 years
  Assessment of cosmetic outcome according to 5-point scoring system
  * Week 1, 2; Month 2, 6, 12, 24, 36, 48, 60
  * At yearly follow-up (photodocumentation in standardized positions) for 5 years
Recurrence Assessment | 5 years
  Recurrence is assessed at month 6, 12, 24, 36, 48, 60

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Wagman, M.D., Study Chair — St. Joseph Hospital of Orange
Locations (1):
- St. Joseph Hospital of Orange, Orange, California, United States